CLINICAL TRIAL: NCT06031025
Title: Prospective Assessment of the Prevalence and Natural History of Gastroesophageal Reflux and Functional Gastro-intestinal Disorders Among At-risk Infants
Brief Title: Prevalence and Natural History of Functional Gastrointestinal Disorders Among At-risk Infants.
Acronym: FUSID
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4921
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Functional Gastrointestinal Disorders; Gastroesophageal Reflux; Constipation - Functional; Diarrhea; Dyschezia; Colic, Infantile; Vomiting; Cyclical
MeSH Terms: conditions — Gastrointestinal Diseases; Gastroesophageal Reflux; Diarrhea; Constipation; Colic; Familial cyclic vomiting syndrome | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire, clinical examination — At each follow up visit, a clinical examination and anthropometric evaluation will be performed. Parents will fill a structured questionnaire to describe the occurrence and characteristics of functional gastrointestinal disorders.

SUMMARY:
The goal of this observational study is to learn about the prevalence and characteristics of functional gastrointestinal disorders (FGID) in at risk infants (former preterm infants and those with birth asphyxia) during the first 2 years of life. The main questions it aims to answer are:

* evaluate the prevalence of symptoms related to gastro-esophageal reflux (GER), of functional gastrointestinal disorders during the first 2 years of life
* describe growth parameters during follow-up up to the corrected age of 2 years Participants will be assessed clinically and with a structured questionnaire based on the Rome IV criteria to describe FGID.

DETAILED DESCRIPTION:
Infants will undergo clinical assessment at 3, 6, 12, 24 months' corrected age at the local Follow-up clinic.

Clinical examination, anthropometric measurement and data from a structured questionnaire to detect FGID will be performed.

Z-scores for weight, length and head circumference will be calculated according to the World Health Organization (WHO) standards.

Data from the questionnaires will be collected. Clinical characteristics of patients and perinatal data will be collected and analyzed by appropriate statistical methods.

The prevalence and characteristics of FGID in the study population will be compared to published data (mostly from term infants).

ELIGIBILITY:
Inclusion Criteria:

* infants with gestational age at birth < 31 weeks
* infants with gestational age at birth < 37 weeks and major respiratory or neurologic morbidity
* infants with history of perinatal asphyxia

Exclusion Criteria:

* lack of informed consent
* diagnosis of congenital or other major gastrointestinal disease (i.e. inflammatory bowel disease, cancer)

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants matching the inclusion criteria will be enrolled in the local Follow-up program (as per clinical routine of the local Institution).
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of FGID | 3, 6, 12, 24 months of corrected age
  Occurrence of FGID (percentage of patients)
Frequency of FGID | 3, 6, 12, 24 months of corrected age
  Frequency of FGID (i.e. number of symptoms per day)
Severity of FGID | 3, 6, 12, 24 months of corrected age
  Severity (scales from 0 to 10 for increasing values) of FGID

SECONDARY OUTCOMES:
Somatic growth: weight | 3, 6, 12, 24 months of corrected age
  Measurement of weight and calculation of z-scores based on reference standards by the World Health Organization
Somatic growth: head circumference | 3, 6, 12, 24 months of corrected age
  Measurement of head circumference and calculation of z-scores based on reference standards by the World Health Organization
Somatic growth: length | 3, 6, 12, 24 months of corrected age
  Measurement of length and calculation of z-scores based on reference standards by the World Health Organization

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nobile, MD, PhD, MSc, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Steutel NF, Zeevenhooven J, Scarpato E, Vandenplas Y, Tabbers MM, Staiano A, Benninga MA. Prevalence of Functional Gastrointestinal Disorders in European Infants and Toddlers. J Pediatr. 2020 Jun;221:107-114. doi: 10.1016/j.jpeds.2020.02.076. PMID 32446468
- [Result] Robin SG, Keller C, Zwiener R, Hyman PE, Nurko S, Saps M, Di Lorenzo C, Shulman RJ, Hyams JS, Palsson O, van Tilburg MAL. Prevalence of Pediatric Functional Gastrointestinal Disorders Utilizing the Rome IV Criteria. J Pediatr. 2018 Apr;195:134-139. doi: 10.1016/j.jpeds.2017.12.012. Epub 2018 Feb 3. PMID 29398057
- [Result] Benninga MA, Faure C, Hyman PE, St James Roberts I, Schechter NL, Nurko S. Childhood Functional Gastrointestinal Disorders: Neonate/Toddler. Gastroenterology. 2016 Feb 15:S0016-5085(16)00182-7. doi: 10.1053/j.gastro.2016.02.016. Online ahead of print. PMID 27144631
- [Result] Iacono G, Merolla R, D'Amico D, Bonci E, Cavataio F, Di Prima L, Scalici C, Indinnimeo L, Averna MR, Carroccio A; Paediatric Study Group on Gastrointestinal Symptoms in Infancy. Gastrointestinal symptoms in infancy: a population-based prospective study. Dig Liver Dis. 2005 Jun;37(6):432-8. doi: 10.1016/j.dld.2005.01.009. Epub 2005 Mar 2. PMID 15893282
- [Result] Scarpato E, Salvatore S, Romano C, Bruzzese D, Ferrara D, Inferrera R, Zeevenhooven J, Steutel NF, Benninga MA, Staiano A. Prevalence and Risk Factors of Functional Gastrointestinal Disorders: A Cross-Sectional Study in Italian Infants and Young Children. J Pediatr Gastroenterol Nutr. 2023 Feb 1;76(2):e27-e35. doi: 10.1097/MPG.0000000000003653. Epub 2022 Nov 1. PMID 36705695